CLINICAL TRIAL: NCT00474357
Title: Myths About Bipolar Affective Disorder: The Role of Structured Group Psychoeducation Therapy
Acronym: BAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lev-Hasharon Mental Healtlh Center (Other Government)
Responsible Party: Dr. Deby Peres, Lev Hasharon Mental Health Center
Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LH55/2007.CTIL
Record Dates: First submitted 2007-05-15; First posted 2007-05-16 (Estimated); Last update posted 2010-12-17 (Estimated); Status verified 2008-05

CONDITIONS: Bipolar Affective Disorder
Keywords: Bipolar affective disorder; myths; preconceived notions; stigma; hope
MeSH Terms: conditions — Bipolar Disorder; Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Bipolar patients participating in psychoeducation intervention
  Interventions: Behavioral: Brief Structured Psychoeducation Group Therapy
- 2 (No Intervention): bipolar patients who do not participate in psychoeducation group
- 3 (No Intervention): Therapists will complete questionnaires regarding myths about bipolar patients, no intervention

INTERVENTIONS:
Behavioral: Brief Structured Psychoeducation Group Therapy — weekly brief structured psychoeducation group therapy for seven weeks for bipolar patients
  Arms: 1

SUMMARY:
This study will examine:

1) The impact of psycho education group therapy sessions relating to beliefs/myths associated with bipolar affective disorder (BAD) on the emotional wellbeing, clinical course and cognition of individuals diagnosed with BAD 2) Will examine the existence of those same beliefs among the various caregivers - psychiatrists, general practitioners, social workers, and psychiatric nurses.

The investigators hypothesize that psychoeducation group therapy will be effective in refuting the myths and will lead to better treatment adherence, longer remissions, fewer hospitalizations, improved self esteem, increased optimism, and better control over the disease process. The investigators also believe that they will identify some beliefs/myths or preconceived notions that are common to both caregivers and individuals with BAD.

DETAILED DESCRIPTION:
Methods:

Effect psychoeducation:

Study population - 30 patients diagnosed with BAD treated in the outpatient clinic, in a state of remission will be evaluated with the Hamilton Rating Scale for Depression, Young Mania Rating Scale, and will then participate in 7 weekly sessions of brief structured psycho education therapy Control group - 30 patients diagnosed with BAD treated in the outpatient clinic, in a state of remission will be evaluated with the Hamilton Rating Scale for Depression, Young Mania Rating Scale. In addition both groups will complete the Snyder Hope Scale, Accepting the Mental Illness Label Scale and a questionnaire regarding Myths in BAD prior to the study, and when the study group finishes their group therapy sessions. (Controls will not participate in the psychoeducation group therapy).

Caregivers beliefs:

50 caregivers from various professions will complete the questionnaire regarding the myths, once only.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of BAD
* State of remission

Exclusion Criteria:

* HAM-D score < 10
* YMRS score < 12
* Has a guardian for either self or property

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-10 (Estimated); Study Completion 2008-10 (Estimated)

PRIMARY OUTCOMES:
Accepting Mental Illness Scale | 7 weeks

SECONDARY OUTCOMES:
Hope Scale | 7 weeks
Myths about BAD questionnaire | 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Igor Oyffe, MD, Study Director — Lev HaSharon Mental Health Center; Deby Peres, MD, Principal Investigator — Lev HaSharon Mental Health Center
Locations (1):
- Lev Hasharon Mental Health Center, Netanya, Israel

REFERENCES:
- See also: Lev-Hasharon Mental Health Center — http://www.lev-hasharon.co.il